CLINICAL TRIAL: NCT04855734
Title: Palliative Care Needs of Children With Rare Diseases and Their Families
Brief Title: FACE for Children With Rare Diseases
Acronym: FACE-Rare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Respecting Choices (Unknown); National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Maureen Lyon, Dr. Maureen Lyon, Ph.D, ABPP, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 00008808; 1R21NR019340-01 (NIH)
Record Dates: First submitted 2021-02-22; First posted 2021-04-22 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Rare Diseases
Keywords: palliative care; psychosocial interventions; rare diseases; family interventions; family-centered care; patient-centered care; pediatrics; adolescent; end-of-life care; public health; mental health; spirituality; children with rare diseases; behavioral interventions; decisional burden; role stress; family caregiver; person-centered care; chronic conditions; complex health needs; caregiver burden; respecting choices; evidence-based practice; randomized clinical trial (RCT); anxiety
MeSH Terms: conditions — Rare Diseases; Psychological Well-Being; Chronic Disease; Caregiver Burden; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Investigators propose a pilot, two-arm, intent-to-treat, single-blinded, single-site, controlled RCT. Family/child dyads (N=30) will be enrolled and randomized to either the FACE-Rare intervention or treatment as usual (TAU) at a 1:1 ratio.
Who Masked: Outcomes Assessor
Masking Description: Study arm allocation will be concealed from the Research Assistant (RA) Assessor to prevent bias during the administration of outcome questionnaires, process measures, and chart abstraction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FACE-Rare Intervention (Experimental): FACE-Rare is a behavioral intervention that combines the CSNAT Pediatric Approach and the Respecting Choices® Next Steps ACP over 3 sessions.
  Sessions 1&2: CSNAT is an evidence-based process of family caregiver assessment and support in specialized medical (palliative) care. The CSNAT tool is structured around 16 categories of family caregiver support. With the goal to decrease caregiver burden, this process consists of 5 stages wherein a nurse or practitioner works with the caregiver to create a shared support plan for the child.
  Session 3: Respecting Choices® Next Steps- This advanced care planning (pACP) conversation engages families in a process for how to make future medical decisions consistent with their goals and values. The interview is structured in 6 stages to achieve 2 main goals: to facilitate conversations with the family about their child's medical condition, history, fears, values, beliefs, and hopes; and to set the stage for the family's future healthcare decisions.
  Interventions: Behavioral: FAmily CEntered (FACE) pACP Intervention
- Treatment-as-Usual (TAU) Control (No Intervention): To minimize the burden to families, we have chosen a Treatment-as-Usual (TAU) comparison condition, where patients will receive their normal standard of care. Both study arms will receive palliative (specialized medical) care information at enrollment and complete questionnaires before and after the intervention or TAU period. Current practice for minors with life-limiting illnesses is to defer initial discussions of advanced care planning (pACP) until a medical crisis, so this is what the TAU control arm condition will consist of.

INTERVENTIONS:
Behavioral: FAmily CEntered (FACE) pACP Intervention — The (approximately) weekly 3-session FACE-Rare intervention of approximately 45-60 minutes each is comprised of the CSNAT approach [Sessions 1 & 2] and Respecting Choices [Session 3].
  Other Names: FACE-Rare Intervention
  Arms: FACE-Rare Intervention

SUMMARY:
Children with ultra-rare or complex rare diseases are routinely excluded from research studies because of their conditions, creating a health disparity. However, new statistical techniques make it possible to study small samples of heterogeneous populations. We propose to study the palliative care needs of family caregivers of children with ultra-rare diseases and to pilot test a palliative care needs assessment and advance care planning intervention to facilitate discussions about the future medical care choices families are likely to be asked to make for their child.

DETAILED DESCRIPTION:
A rare disease is a condition affecting fewer than 200,000 persons. Pediatric patients with rare diseases experience high mortality with 30% not living to see their 5th birthday. Families are likely to be asked to make complex medical decisions for their child. Pediatric advance care planning involves preparation and skill development to help make future medical care choices. Children with rare disorders are a heterogeneous group often with co-morbidities, resulting in their exclusion from research, thereby creating a health disparity for this vulnerable population. Available research on families of children with rare diseases lacks scientific rigor. Although desperately needed, there are few empirically validated interventions to address these issues. We propose to close a gap in our knowledge of families' needs for support in a heterogeneous group of children with rare diseases; and to test an advance care planning intervention.

The FAmily CEntered (FACE) pediatric advance care planning intervention, proven successful with cancer and HIV, is adapted to families with children who have rare diseases. Theoretically informed and developed by the PI, Dr. Lyon, and colleagues, the proposed intervention will use Respecting Choices Next Steps Pediatric Advance Care Planning™ for families whose child is unable to participate in health care decision-making. Our consultation with families of children with rare disorders and the National Organization for Rare Disorders (NORD) revealed that basic palliative care needs should be addressed first, before an advance care planning intervention. For the study to be able to meet this request, all families randomized to the intervention will first complete the Carer Support Needs Assessment Tool (CSNAT)© which our investigative team adapted for use in pediatrics. In the CSNAT Approach, facilitators assess caregivers' prioritized palliative care needs and develop Shared Action Plans for palliative care support. Thus, we propose an innovative 3-session FACE-Rare intervention, integrating two evidence-based approaches. We will evaluate FACE-Rare using a scientifically rigorous intent-to-treat, single-blinded, randomized controlled trial design. Family/child pairs or dyads (N=30 dyads) will be randomized to FACE-Rare (CSNAT Sessions 1 & 2 plus Respecting Choices Sessions 3) or control (Treatment As Usual) groups. Both groups will receive palliative care information. All families will complete questionnaires at baseline and 3-months follow-up. Investigators will evaluate the initial efficacy of FACE-Rare on family quality of life (psychological, spiritual). We will estimate how religiousness and caregiver appraisal influence families' quality of life. We will also explore health care utilization by the children during the study and family satisfaction.

If the aims of this pilot trial are achieved, a future, large, multi-site trial will test the full theoretical model to improve care for children with rare diseases and their families through family engaged pediatric Advance Care Planning. The ultimate goal is to minimize suffering and enhance the quality of life of family caregivers of children with rare diseases; and through this process to improve the palliative care of their children.

ELIGIBILITY:
Inclusion Criteria:

Child inclusion criteria are

1. ≥1.0 years and <18.0 years at enrollment;e
2. unable to participate in end-of-life care decision-making;
3. have a rare disease as operationally defined (See Human Subjects);
4. not under a Do Not Resuscitate Order or Allow a Natural Death Order; and
5. not in the Intensive Care Unit.

Family caregiver inclusion criteria are:

1. ≥ 18.0 years at enrollment;
2. legal guardian of child and child's caregiver;
3. can speak and understand English; and
4. not known to be developmentally delayed.

Exclusion Criteria:

(1) Family caregiver is actively homicidal, suicidal, or psychotic at the time of enrollment.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen E Lyon, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
The proposed research will include data from 30 children living with rare diseases who are unable to participate in their own medical care decision-making and their 30 family caregivers. The final dataset will be stripped of individual-level identifiable data prior to release for sharing. Given the vulnerable nature of the subjects (child participants), we will make the data and associated documentation available to researchers under a data-sharing agreement that includes:
  1. appropriate human-subjects review and approval; and
  2. a commitment to use the data only for research purposes and that no attempt will be made to identify individual participants.
  The Biostatistics group will perform the mechanics of de-identification and provide the data in an agreed-upon format. De-identification will include stripping the data of PHI; removing dates or adding a random offset to the dates. Only de-identified group data will be shared. This protects participant confidentiality.

REFERENCES:
- [Background] Lyon ME, Wiener L. Special Issue: Psychosocial Considerations for Children and Adolescents Living with a Rare Disease. Children (Basel). 2022 Jul 21;9(7):1099. doi: 10.3390/children9071099. PMID 35884083
- [Background] Sandquist M, Davenport T, Monaco J, Lyon ME. The Transition to Adulthood for Youth Living with Rare Diseases. Children (Basel). 2022 May 12;9(5):710. doi: 10.3390/children9050710. PMID 35626888
- [Background] Fratantoni K, Livingston J, Schellinger SE, Aoun SM, Lyon ME. Family-Centered Advance Care Planning: What Matters Most for Parents of Children with Rare Diseases. Children (Basel). 2022 Mar 21;9(3):445. doi: 10.3390/children9030445. PMID 35327817
- [Background] Aoun SM, Stegmann R, Deleuil R, Momber S, Cuddeford L, Phillips MB, Lyon ME, Gill FJ. "It Is a Whole Different Life from the Life I Used to Live": Assessing Parents' Support Needs in Paediatric Palliative Care. Children (Basel). 2022 Mar 1;9(3):322. doi: 10.3390/children9030322. PMID 35327694
- [Background] Lyon ME, Thompkins JD, Fratantoni K, Fraser JL, Schellinger SE, Briggs L, Friebert S, Aoun S, Cheng YI, Wang J. Family caregivers of children and adolescents with rare diseases: a novel palliative care intervention. BMJ Support Palliat Care. 2022 Nov;12(e5):e705-e714. doi: 10.1136/bmjspcare-2019-001766. Epub 2019 Jul 25. PMID 31345846
- [Background] Aoun SM, Gill FJ, Phillips MB, Momber S, Cuddeford L, Deleuil R, Stegmann R, Howting D, Lyon ME. The profile and support needs of parents in paediatric palliative care: comparing cancer and non-cancer groups. Palliat Care Soc Pract. 2020 Sep 25;14:2632352420958000. doi: 10.1177/2632352420958000. eCollection 2020. PMID 33033802
- [Result] - Kreicbergs U (Discussant), Handberg C, Udo C, Thompkins J (presenter) Lyon ME (organizer). Symposium: Lessons Learned during the COVID-19 and Beyond Pandemic for Children Living with Rare Diseases and their Siblings. Lyon Presentation: Family Identified Palliative Care Needs of FAmily Caregivers of Children Living with Rare Diseases during COVID-19-United States 7th Public Health Palliative Care International Conference. September 21, 2022. Bruges, Belgium.
- [Result] - Lyon, ME, Fraser J, Thompkins J (presenter). FACE Rare: A novel palliative care intervention for family caregivers of children and adolescents living with a rare disease. Podium Presentation. University of Pittsburgh's National Center on Family Support's Second Biennial Conference on Caregiving Research. Building Bridges: Advancing Family Caregiving Research Across the Lifespan, National Center on Caregiving. Pittsburg, PA. October 1, 2022.
- [Result] Lyon ML. Detwiler K, Torres C, Guerrera MF, Thompkins J. FACE-Rare: A Novel Intervention for Family Caregivers of Children Living with Rare Diseases. BMJ Supportive & Palliative Care 2023;13(Suppl 4):A16.
- See also: Lyon ML. Detwiler K, Torres C, Guerrera MF, Thompkins J. FACE-Rare: A Novel Intervention for Family Caregivers of Children Living with Rare Diseases. BMJ Supportive & Palliative Care 2023;13(Suppl 4):A16. — https://doi.org/10.1136/spcare-2023-ACP.39

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Family caregivers were recruited from outpatient clinics at Children's National Hospital, a quaternary pediatric hospital. There were 21 children and 21 primary family caregivers enrolled in the study. Randomization was at the level of the dyad (child with a rare disease and the primary family caregiver). Thus, 42 participants (21 child/family dyads) completed the baseline assessment and were then randomized. The flow chart is reported as adolescent/family dyads.
Groups:
- FACE-Rare Intervention: FACE-Rare is a behavioral intervention that combines the CSNAT Pediatric Approach and the Respecting Choices® Next Steps ACP over 3 sessions.
  Sessions 1&2: CSNAT is an evidence-based process of family caregiver assessment and support in specialized medical (palliative) care. The CSNAT tool is structured around 16 categories of family caregiver support. With the goal to decrease caregiver burden, this process consists of 5 stages wherein a nurse or practitioner works with the caregiver to create a shared support plan for the child.
  Session 3: Respecting Choices® Next Steps- This advanced care planning (pACP) conversation engages families in a process for how to make future medical decisions consistent with their goals and values. The interview is structured in 6 stages to achieve 2 main goals: to facilitate conversations with the family about their child's medical condition, history, fears, values, beliefs, and hopes; and to set the stage for the family's future healthcare decisions.
  FAmily CEntered (FACE) pACP Intervention: The (approximately) weekly 3-session FACE-Rare intervention of approximately 45-60 minutes each is comprised of the CSNAT approach [Sessions 1 & 2] and Respecting Choices [Session 3].
Period: Overall Study
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Started (Randomization at a ratio of 1:1. Randomization was at the level of the child/caregiver dyad: 9 dyads in intervention, 12 dyads in TAU.) | 18 (9 child/caregiver dyads) | 24 (12 child/caregiver dyads)
Children | 9 | 12
Caregivers | 9 | 12
Completed (Completed are child/caregiver dyads.) | 16 (8 child/caregiver dyads completed intervention. One child/family dyad was lost to follow-up after randomization but before beginning the 3-session intervention.) | 22 (11 child/caregiver dyads completed TAU. One child/family dyad completed the process measures at 3 weeks post-baseline but was lost to 3-month follow-up.)
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: 42 participants (21 child with rare disease and child's primary caregiver dyads) completed baseline assessment. Baseline analysis was at level of participant with separate analysis for child with rare disease and family caregiver.
Groups:
- Total: Total of all reporting groups
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control | Total
Number analyzed (Participants) | 18 | 24 | 42
Age, Categorical [Count of Participants; unit: Participants] — Demographic data were collected on a standardized form. Child's age was measured by family caregiver report and family caregiver age was measured by self-report. Population: Baseline analysis was at level of participant with separate analysis for children with rare diseases and the primary family caregiver.
  Participants
    Child with rare disease: number analyzed (Participants) | 9 | 12 | 21
    Child with rare disease: <=18 years | 9 | 12 | 21
    Child with rare disease: Between 18 and 65 years | 0 | 0 | 0
    Child with rare disease: >=65 years | 0 | 0 | 0
    Primary family caregiver: number analyzed (Participants) | 9 | 12 | 21
    Primary family caregiver: <=18 years | 0 | 0 | 0
    Primary family caregiver: Between 18 and 65 years | 9 | 12 | 21
    Primary family caregiver: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Demographic information was collected on a standardized form. Sex of child was based on child's family caregiver report. Sex of primary family caregiver was based on primary family caregiver self-report. Population: Sex as a biological variable was analyzed as a separate variable for child and primary family caregiver.
  Participants
    Child with rare disease: number analyzed (Participants) | 9 | 12 | 21
    Child with rare disease: Female | 5 | 6 | 11
    Child with rare disease: Male | 4 | 6 | 10
    Primary family caregiver: number analyzed (Participants) | 9 | 12 | 21
    Primary family caregiver: Female | 7 | 10 | 17
    Primary family caregiver: Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Demographic data were collected on a standardized form. Child's race was reported by family caregiver. Family caregiver's race was self-reported. Population: Analysis of the population was at the level of the individual and not the dyad. We analyzed separately age data for child from age data for primary family caregiver.
  Participants
    Child with rare disease: number analyzed (Participants) | 9 | 12 | 21
    Child with rare disease: American Indian or Alaska Native | 0 | 0 | 0
    Child with rare disease: Asian | 0 | 0 | 0
    Child with rare disease: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Child with rare disease: Black or African American | 4 | 1 | 5
    Child with rare disease: White | 3 | 10 | 13
    Child with rare disease: More than one race | 2 | 1 | 3
    Child with rare disease: Unknown or Not Reported | 0 | 0 | 0
    Primary family caregiver: number analyzed (Participants) | 9 | 12 | 21
    Primary family caregiver: American Indian or Alaska Native | 0 | 0 | 0
    Primary family caregiver: Asian | 0 | 0 | 0
    Primary family caregiver: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Primary family caregiver: Black or African American | 3 | 1 | 4
    Primary family caregiver: White | 5 | 10 | 15
    Primary family caregiver: More than one race | 1 | 1 | 2
    Primary family caregiver: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — All participants were recruited from Children's National Hospital in Washington, DC, in the United States of America. No additional details, such as zip code, were collected from participants.
  participants
    United States | 18 | 24 | 42

OUTCOME MEASURES:

1. Primary Outcome: Beck Anxiety Inventory
Description: The Beck Anxiety Inventory (BAI) is a 21-item measure of anxiety rated on a 4-point Likert scale of symptoms over the past week. The BAI has demonstrated reliability and validity to assess anxiety in individuals aged 17-80 years. The BAI has good reliability and validity for family caregivers of seriously ill children. It is a measure of Quality of life: emotional health. Higher scores mean more anxiety symptoms. Total score was used in analysis. Scores range from 0-63.
Time Frame: Change from Baseline Anxiety at 3 Months Post-Enrollment
Population: Data analysis was with the family caregivers.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 9 | 12
score on a scale
  Baseline Total score | 10.4 (8.5) | 9.5 (9.5)
  3 month follow-up Total Score | 11.1 (8.0) | 8.5 (9.6)
Statistical Analysis 1: Comparison: FACE-Rare Intervention vs Treatment-as-Usual (TAU) Control; Test type: Superiority; p = 0.835, Mixed Models Analysis — Threshold for significance was <0.05; Mean ratio = 0.962, 95% CI 2-sided [0.661 to 1.396]

2. Primary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)- Spiritual Well-Being Scale, Version 4
Description: Assessed construct of spiritual well-being. Two subscales Meaning/Peace (7 items) and Faith (5 items) and Total score (12 items) were calculated. on a 5-point Likert scale from 0=not at all to 5=very much. Some items are reverse scored. See www.facit.org Meaning/Peace subscale score range from minimum value of 0 to maximum value of 32. Higher scores indicate better meaning/peace. Faith subscale score range from 0 minimum value to maximum value of 16. Higher scores indicate better meaning/peace. Higher scores indicate better spiritual well-being.
Time Frame: Change from Baseline Spiritual Well-Being at 3 Months Post-Enrollment
Population: Family caregivers of children with rare diseases.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 9 | 12
score on a scale
  Baseline Meaning/Peace | 24.0 [23.0 to 27.0] | 25.0 [23.5 to 27.0]
  3 month Meaning/Peace | 26.0 [24.0 to 30.0] | 26.0 [21.8 to 29.0]
  Baseline Faith | 11.0 [10.0 to 14.0] | 6.0 [3.8 to 7.5]
  3 month Faith | 9.0 [7.0 to 14.0] | 7.0 [4.8 to 11.0]
Statistical Analysis 1: Comparison: FACE-Rare Intervention vs Treatment-as-Usual (TAU) Control; Meaning/Peace subscale which was a primary outcome; Test type: Superiority; p = 0.032, Mixed Models Analysis — <0.05 was threshold for significance level; Mean ratio = 0.826, 95% CI 2-sided [0.75 to 0.986]

3. Primary Outcome: Advance Care Plan Document for Children With Rare Diseases
Description: Advanced Care Planning (ACP) Documentation in Electronic Health Records (EHR). Score will be present in EHR or absent from EHR. Evidence of any advance care document (yes/no) will count.
Time Frame: Change from Baseline ACP Documentation in the Electronic Health Record at 12 weeks Post-Enrollment
Population: Advance care plan for child documented in the Electronic Health Record.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 9 | 12
Participants
  Baseline: No | 8 | 12
  Baseline: Yes | 1 | 0
  3-month follow-up: No | 6 | 12
  3-month follow-up: Yes | 3 | 0

4. Primary Outcome: Days in Palliative Care Prior to Death
Description: Score is number of days patient was enrolled in a palliative care program in the 30 days prior to death. Applicable only to patients who have deceased since study enrollment. Used to standardize child healthcare utilization from data abstraction based on retrospective medical chart review. Minimum value is 0 with no maximum. Higher score indicates higher level of healthcare utilization.
Time Frame: 12 weeks Post-Enrollment
Population: Child with rare disease. No child with a rare disease died during the study, so data for Days in Palliative Care Prior to death was not collected.
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Hospitalizations
Description: Used to standardize child healthcare utilization from data abstraction by the research nurse based on medical chart review in Electronic Health Record. Score is recorded number of inpatient hospital admissions for clinical treatment for the child with a rare disease. Minimum value is 0 with no maximum. Higher score indicates higher level of healthcare utilization. Questions was "Hospitalization in the last 3 months?"
Time Frame: Change from Baseline to Frequency at 12 weeks Post-Enrollment
Population: Children with rare diseases.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 9 | 12
Participants
  Baseline: No | 7 | 7
  Baseline: Yes | 2 | 5
  3-month follow-up: No | 7 | 8
  3-month follow-up: Yes | 2 | 4

6. Primary Outcome: Place of Death
Description: Location where the patient was pronounced dead, as reported in their EMR. Applicable only to patients who have deceased since study enrollment. Categories are Inpatient hospice setting, Home with hospice, Home without hospice, Hospital ICU, Hospital-Not ICU, Other, or Unknown. Used to standardize child healthcare utilization from data abstraction based on retrospective medical chart review.
Time Frame: 12 weeks Post-Enrollment
Population: Child with a rare disease. No child with a rare disease died during the study, so Place of Death was not collected.
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Brief-Multidimensional Measure of Religion and Spirituality - Responses to Question 1
Description: Survey responses to: 1. How often do you feel God's presence? On 6-point Likert-scale responses range from every day to never or almost never.
Time Frame: Baseline and 3-month follow-up.
Population: Primary family caregivers of children with rare diseases.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 9 | 12
Participants
  Baseline How often do you feel God's presence?: Declined | 1 | 0
  Baseline How often do you feel God's presence?: Every day | 3 | 1
  Baseline How often do you feel God's presence?: Most days | 1 | 3
  Baseline How often do you feel God's presence?: Once in a while | 3 | 5
  Baseline How often do you feel God's presence?: Some days | 1 | 2
  Baseline How often do you feel God's presence?: Many times a day. | 0 | 0
  Baseline How often do you feel God's presence?: Never or almost never | 0 | 1
  3-month follow up -How often do you feel God's presence?: Declined | 0 | 0
  3-month follow up -How often do you feel God's presence?: Every day | 2 | 4
  3-month follow up -How often do you feel God's presence?: Most days | 2 | 2
  3-month follow up -How often do you feel God's presence?: Once in a while | 1 | 5
  3-month follow up -How often do you feel God's presence?: Some days | 1 | 0
  3-month follow up -How often do you feel God's presence?: Many times a day. | 1 | 1
  3-month follow up -How often do you feel God's presence?: Never or almost never | 2 | 0

8. Secondary Outcome: Family Appraisal of Caregiving Questionnaire for Palliative Care for Palliative Care (FACQ-PC)
Description: The FACQ-PC is a 25-item measure consists of four theoretically derived subscales: (i) caregiver strain, (ii) positive caregiving appraisals, (iii) caregiver distress, and (iv) family well-being. Scores are from 5 = strongly agree to 1 = strongly disagree. We did not calculate a Total score. We only used the 4 subscale scores. On the subscale scores for positive caregiving appraisals and family well-being, higher scores mean better outcomes, i.e. greater positive caregiving appraisals or family well-being. On the subscale scores for caregiver strain and caregiver distress, higher scores mean worse outcomes, i.e. greater caregiver strain or caregiver distress. The FACQ-PC subscale scores were computed by taking the mean of the items (score range 1-5). Some items were reverse scored, depending on how the item is phrased, so that higher scores = higher amount of the subscale being measured. So the minimum value for each subscale is 1 and the maximum value for each subscale is 5.
Time Frame: Change from Baseline appraisal of Caregiving at 12 weeks Post-Enrollment
Population: Primary family caregivers of children with a rare disease.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 9 | 12
score on a scale
  Caregiver strain subscale baseline | 3.3 [2.9 to 3.6] | 3.0 [2.4 to 3.7]
  Positive caregiving appraisals Baseline | 4.7 [4.1 to 4.9] | 4.6 [4.3 to 4.7]
  Caregiver Distress Baseline | 3.3 [2.8 to 3.8] | 3.5 [2.9 to 4.0]
  Family well-being baseline | 4.2 [3.5 to 4.7] | 4.2 [3.9 to 4.5]
  caregiver strain 3 Month follow up | 3.5 [2.8 to 3.8] | 2.9 [2.5 to 3.9]
  Positive caregiving appraisals 3 month follow up | 4.7 [4.3 to 5.0] | 4.6 [4.5 to 4.9]
  Caregiver distress 3 month follow up | 2.8 [2.5 to 3.3] | 3.4 [2.3 to 3.8]
  Family well-being 3 month follow up | 4.5 [3.8 to 4.5] | 4.2 [4.0 to 4.4]
Statistical Analysis 1: Comparison: FACE-Rare Intervention vs Treatment-as-Usual (TAU) Control; Caregiver strain subscale scores at 3 months post-intervention comparing intervention to TAU, controlling for baseline levels; Test type: Superiority; p = 0.284, Mixed Models Analysis — <0.05 threshold for significance level; Mean ratio = 1.052, 95% CI 2-sided [0.959 to 1.157]
Statistical Analysis 2: Comparison: FACE-Rare Intervention vs Treatment-as-Usual (TAU) Control; Caregiver distress subscale controlling for baseline levels; Test type: Superiority; p = 0.228, Mixed Models Analysis — <0.05 threshold for significance level; Mean ratioj = 0.931, 95% CI 2-sided [0.827 to 1.048]
Statistical Analysis 3: Comparison: FACE-Rare Intervention vs Treatment-as-Usual (TAU) Control; Family well-being subscale controlling for baseline levels; Test type: Superiority; p = 0.504, Mixed Models Analysis — <0.05 significance level; Mean ratio = 0.984, 95% CI 2-sided [0.94 to 1.032]
Statistical Analysis 4: Comparison: FACE-Rare Intervention vs Treatment-as-Usual (TAU) Control; Positive Caregiving Appraisals subscale at 3 month follow up, controlling for baseline levels; Test type: Superiority; p = 0.741, Mixed Models Analysis — <0.05 significance level; Mean ratio = 0.995, 95% CI 2-sided [0.967 to 1.024]

9. Secondary Outcome: Hickman Role Stress Decisional Burden Scale
Description: Visual analogue scale 0-100. "How stressful is it for you to make medical decisions for your child?" 1 item. Higher score means more stress, lower scores mean less stress.
Time Frame: Up to 5 Weeks Post-Enrollment
Population: Primary caregiver of child with rare disease.
Measure: Median (Inter-Quartile Range); unit: raw score units on a scale
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 9 | 12
raw score units on a scale
  Baseline | 75 [47.0 to 90.0] | 71.0 [39.3 to 88.0]
  3-month follow-up | 75.0 [75.0 to 85.0] | 72.5 [50.0 to 81.3]

10. Secondary Outcome: Brief Multidimensional Measurement of Religiousness/Spirituality (BMMRS-adapted) Survey Responses to Question 2.
Description: Responses to survey question 2, How often do you pray privately? 7 point Likert scale ranging from a few times a month to once a day. Higher scores in pray item indicate more prayer.
Time Frame: Baseline and 3-month follow-up
Population: Family caregivers of children with rare diseases.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 9 | 12
Participants
  Baseline How often do you pray privately?: A few times a month | 2 | 2
  Baseline How often do you pray privately?: A few times a week | 1 | 3
  Baseline How often do you pray privately?: More than once a day | 3 | 3
  Baseline How often do you pray privately?: Never | 1 | 2
  Baseline How often do you pray privately?: Once a month | 2 | 0
  Baseline How often do you pray privately?: Less than once a month | 0 | 1
  Baseline How often do you pray privately?: Once a day | 0 | 1
  3 month follow-up How often do you pray privately?: A few times a month | 2 | 2
  3 month follow-up How often do you pray privately?: A few times a week | 2 | 4
  3 month follow-up How often do you pray privately?: More than once a day | 3 | 3
  3 month follow-up How often do you pray privately?: Never | 1 | 1
  3 month follow-up How often do you pray privately?: Once a month | 1 | 0
  3 month follow-up How often do you pray privately?: Less than once a month | 0 | 1
  3 month follow-up How often do you pray privately?: Once a day | 0 | 1

11. Other Pre Specified Outcome: Satisfaction Questionnaire (Process Measure)
Description: Items for this 13-item assessment of family satisfaction with the intervention were developed using input from the community about the emotional aspects of participation. Items are on a 5-point Likert scale from strongly disagree to strongly agree. 6 items were negative (felt afraid, too much to handle, harmful, angry, sad hurtful) and 7 items were positive (useful, helpful, load off my mind, satisfied, something I needed to do, courageous, worthwhile). Each item was scored separately. Higher score for positive scale was better outcome. Higher score for negative scale was worse outcome. Study-specific process measure to assess adverse events and benefit/burden of participation. 12 items Total.
Time Frame: Up to 5 Weeks Post-Baseline
Population: Family caregivers of children with rare diseases
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 9 | 12
Participants
  1. It was useful: Strongly disagree | 0 | 1
  1. It was useful: Disagree | 0 | 2
  1. It was useful: Neither agree or disagree. | 3 | 4
  1. It was useful: Agree | 3 | 4
  1. It was useful: Strongly agree. | 3 | 1
  2. It was helpful: Strongly disagree | 0 | 1
  2. It was helpful: Disagree | 0 | 2
  2. It was helpful: Neither agree or disagree. | 3 | 4
  2. It was helpful: Agree | 4 | 4
  2. It was helpful: Strongly agree. | 2 | 1
  3. I felt scared or afraid: Strongly disagree | 4 | 9
  3. I felt scared or afraid: Disagree | 3 | 2
  3. I felt scared or afraid: Neither agree or disagree. | 2 | 0
  3. I felt scared or afraid: Agree | 0 | 1
  3. I felt scared or afraid: Strongly agree. | 0 | 0
  4. It felt like a load off my mind.: Strongly disagree | 0 | 1
  4. It felt like a load off my mind.: Disagree | 3 | 3
  4. It felt like a load off my mind.: Neither agree or disagree. | 2 | 7
  4. It felt like a load off my mind.: Agree | 4 | 1
  4. It felt like a load off my mind.: Strongly agree. | 0 | 0
  5. It was too much to handle.: Strongly disagree | 3 | 5
  5. It was too much to handle.: Disagree | 4 | 5
  5. It was too much to handle.: Neither agree or disagree. | 0 | 1
  5. It was too much to handle.: Agree | 2 | 1
  5. It was too much to handle.: Strongly agree. | 0 | 0
  6. I felt satisfied.: Strongly disagree | 0 | 0
  6. I felt satisfied.: Disagree | 1 | 2
  6. I felt satisfied.: Neither agree or disagree. | 2 | 4
  6. I felt satisfied.: Agree | 6 | 4
  6. I felt satisfied.: Strongly agree. | 0 | 2
  7. It was harmful.: Strongly disagree | 6 | 10
  7. It was harmful.: Disagree | 3 | 1
  7. It was harmful.: Neither agree or disagree. | 0 | 1
  7. It was harmful.: Agree | 0 | 0
  7. It was harmful.: Strongly agree. | 0 | 0
  8. I felt angry.: Strongly disagree | 6 | 10
  8. I felt angry.: Disagree | 3 | 1
  8. I felt angry.: Neither agree or disagree. | 0 | 1
  8. I felt angry.: Agree | 0 | 0
  8. I felt angry.: Strongly agree. | 0 | 0
  9. It was something I needed to do.: Strongly disagree | 0 | 1
  9. It was something I needed to do.: Disagree | 1 | 0
  9. It was something I needed to do.: Neither agree or disagree. | 1 | 5
  9. It was something I needed to do.: Agree | 4 | 4
  9. It was something I needed to do.: Strongly agree. | 3 | 2
  10. I felt sad.: Strongly disagree | 1 | 7
  10. I felt sad.: Disagree | 2 | 3
  10. I felt sad.: Neither agree or disagree. | 0 | 1
  10. I felt sad.: Agree | 5 | 1
  10. I felt sad.: Strongly agree. | 1 | 0
  111. I felt courageous.: Strongly disagree | 1 | 1
  111. I felt courageous.: Disagree | 2 | 2
  111. I felt courageous.: Neither agree or disagree. | 3 | 6
  111. I felt courageous.: Agree | 3 | 1
  111. I felt courageous.: Strongly agree. | 0 | 2
  12. It felt harmful.: Strongly disagree | 5 | 9
  12. It felt harmful.: Disagree | 4 | 1
  12. It felt harmful.: Neither agree or disagree. | 0 | 2
  12. It felt harmful.: Agree | 0 | 0
  12. It felt harmful.: Strongly agree. | 0 | 0
  13. It was worthwhile.: Strongly disagree | 0 | 1
  13. It was worthwhile.: Disagree | 0 | 0
  13. It was worthwhile.: Neither agree or disagree. | 0 | 2
  13. It was worthwhile.: Agree | 7 | 7
  13. It was worthwhile.: Strongly agree. | 2 | 2

12. Other Pre Specified Outcome: Quality of Communication Questionnaire
Description: This is a process, not an outcome, measure. The participant is asked to rate how good the facilitator was for each of 4 communication skills on a scale from 0, definitely no, to 5, definitely yes. Higher scores mean better communication. Minimum score was 4. Maximum score was 20. We did not calculate a total score, as this was a process measure to assess the facilitator's communication and to provide feedback to the facilitator.
Time Frame: Up to 5 Weeks Post-Baseline
Population: Family caregivers of children living with rare diseases.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 9 | 12
Participants
  1. Do you think that your attitudes are known by the interviewer?: Definitely yes | 4 | 1
  1. Do you think that your attitudes are known by the interviewer?: Do Not Know | 1 | 5
  1. Do you think that your attitudes are known by the interviewer?: Probably yes | 4 | 3
  1. Do you think that your attitudes are known by the interviewer?: Declined | 0 | 1
  1. Do you think that your attitudes are known by the interviewer?: Definitely no | 0 | 1
  1. Do you think that your attitudes are known by the interviewer?: Missing | 0 | 1
  2. Did you feel that the interviewer cared about you as a person?: Definitely yes | 8 | 6
  2. Did you feel that the interviewer cared about you as a person?: Do Not Know | 0 | 1
  2. Did you feel that the interviewer cared about you as a person?: Probably yes | 1 | 3
  2. Did you feel that the interviewer cared about you as a person?: Declined | 0 | 1
  2. Did you feel that the interviewer cared about you as a person?: Definitely no | 0 | 0
  2. Did you feel that the interviewer cared about you as a person?: Missing | 0 | 1
  3. Did you feel that the interviewer listened to what you said?: Definitely yes | 9 | 8
  3. Did you feel that the interviewer listened to what you said?: Do Not Know | 0 | 0
  3. Did you feel that the interviewer listened to what you said?: Probably yes | 0 | 2
  3. Did you feel that the interviewer listened to what you said?: Declined | 0 | 1
  3. Did you feel that the interviewer listened to what you said?: Definitely no | 0 | 0
  3. Did you feel that the interviewer listened to what you said?: Missing | 0 | 1
  4. Did you feel that the interviewer gave you enough attention?: Definitely yes | 9 | 10
  4. Did you feel that the interviewer gave you enough attention?: Do Not Know | 0 | 0
  4. Did you feel that the interviewer gave you enough attention?: Probably yes | 0 | 0
  4. Did you feel that the interviewer gave you enough attention?: Declined | 0 | 1
  4. Did you feel that the interviewer gave you enough attention?: Definitely no | 0 | 0
  4. Did you feel that the interviewer gave you enough attention?: Missing | 0 | 1

13. Other Pre Specified Outcome: Brief Multidimensional Measure of Religiousness/Spirituality (Brief MMRS) "How Often do You go to Religious Services?"
Description: Responses to "How often do you go to religious services?" Responses ranged from "once or twice a year" to "more than once a week." Higher scores indicated greater attendance at religious services. Responses were used as a covariate in the initial Generalized linear mixed effect models. Prior research had indicated that this variable moderated quality of life outcomes. Higher scores indicate more attendance at religious services.
Time Frame: Baseline to 3 month follow-up
Population: Family caregivers of children with rare diseases.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 9 | 12
Participants
  How often do you go to religious services? baseline: Every month or so | 1 | 2
  How often do you go to religious services? baseline: Never | 3 | 3
  How often do you go to religious services? baseline: Once or twice a month | 2 | 1
  How often do you go to religious services? baseline: Once or twice a year | 3 | 3
  How often do you go to religious services? baseline: Every week or more often | 0 | 2
  How often do you go to religious services? baseline: More than once a week | 0 | 1
  How often do you go to religious services? 3 month follow up: Every month or so | 2 | 1
  How often do you go to religious services? 3 month follow up: Never | 3 | 4
  How often do you go to religious services? 3 month follow up: Once or twice a month | 3 | 1
  How often do you go to religious services? 3 month follow up: Once or twice a year | 1 | 3
  How often do you go to religious services? 3 month follow up: Every week or more often | 0 | 3
  How often do you go to religious services? 3 month follow up: More than once a week | 0 | 0

14. Other Pre Specified Outcome: Brief Multidimensional Measure of Religiousness/Spirituality (Brief MMRS): "To What Extent do You Consider Yourself a Religious Person?"
Description: Responses to "To what extent do you consider yourself a religious person?" Responses ranged from "moderately religious" to "not religious at all." Higher scores indicated higher religiousness. Responses were collected as a covariate in the initial Generalized linear mixed effect models. Prior research had indicated that this variable moderated quality of life outcomes. Higher scores in the religious indicate self-perception as a more religious person.
Time Frame: Baseline and 3 month follow-up
Population: Family caregivers of children with rare diseases.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 9 | 12
Participants
  To what extent do you consider yourself a religious person? Baseline: Moderately religious | 3 | 4
  To what extent do you consider yourself a religious person? Baseline: Not religious at all | 3 | 2
  To what extent do you consider yourself a religious person? Baseline: Slightly religious | 1 | 4
  To what extent do you consider yourself a religious person? Baseline: Very religious | 2 | 2
  To what extent do you consider yourself a religious person? 3 month follow up: Moderately religious | 2 | 2
  To what extent do you consider yourself a religious person? 3 month follow up: Not religious at all | 2 | 3
  To what extent do you consider yourself a religious person? 3 month follow up: Slightly religious | 3 | 6
  To what extent do you consider yourself a religious person? 3 month follow up: Very religious | 2 | 1

15. Other Pre Specified Outcome: Brief Multidimensional Measurement of Religiousness/Spirituality (BMMRS-adapted): To What Extent do You Consider Yourself a Spiritual Person?
Description: Responses to "To What Extent do You Consider Yourself a spiritual person?" Responses ranged from "not spiritual at all" to "very spiritual." Higher score meant more spiritual. Reported are frequency distributions and percentages. A higher score on the spiritual person item indicates self-perception as more spiritual.
Time Frame: Baseline to 3 month outcomes.
Population: Family caregivers of children with rare diseases.
Measure: Count of Participants; unit: Participants
Arm/Group | FACE-Rare Intervention | Treatment-as-Usual (TAU) Control
Number analyzed (Participants) | 9 | 12
Participants
  To what extent do you consider yourself a spiritual person? Baseline: Moderately spiritual | 3 | 7
  To what extent do you consider yourself a spiritual person? Baseline: Not spiritual at all | 1 | 0
  To what extent do you consider yourself a spiritual person? Baseline: Slightly spiritual | 2 | 5
  To what extent do you consider yourself a spiritual person? Baseline: Very spiritual | 3 | 0
  To what extent do you consider yourself a spiritual person? 3 month follow up: Moderately spiritual | 2 | 4
  To what extent do you consider yourself a spiritual person? 3 month follow up: Not spiritual at all | 1 | 0
  To what extent do you consider yourself a spiritual person? 3 month follow up: Slightly spiritual | 3 | 4
  To what extent do you consider yourself a spiritual person? 3 month follow up: Very spiritual | 3 | 4

ADVERSE EVENTS:
Time Frame: From enrollment through study completion up to 3 months post-intervention (+/- 1 month study window).
Description: Potential adverse event data were collected over the 2 year trial period and reported to annual meetings with the Safety Monitoring Committee. Weekly team meetings at this single site consistently reviewed potential adverse events, which included review of all study participant interactions. No patients or family caregivers died during the pilot trial.
Groups:
- FACE-Rare Intervention-Children: FACE-Rare is a behavioral intervention that combines the CSNAT Pediatric Approach and the Respecting Choices® Next Steps ACP over 3 sessions.
  Sessions 1&2: CSNAT is an evidence-based process of family caregiver assessment and support in specialized medical (palliative) care. The CSNAT tool is structured around 16 categories of family caregiver support. With the goal to decrease caregiver burden, this process consists of 5 stages wherein a nurse or practitioner works with the caregiver to create a shared support plan for the child.
  Session 3: Respecting Choices® Next Steps- This advanced care planning (pACP) conversation engages families in a process for how to make future medical decisions consistent with their goals and values. The interview is structured in 6 stages to achieve 2 main goals: to facilitate conversations with the family about their child's medical condition, history, fears, values, beliefs, and hopes; and to set the stage for the family's future healthcare decisions.
  FAmily CEntered (FACE) pACP Intervention: The (approximately) weekly 3-session FACE-Rare intervention of approximately 45-60 minutes each is comprised of the CSNAT approach [Sessions 1 & 2] and Respecting Choices [Session 3].
- Treatment-as-Usual (TAU) Control- Children; TAU-control-Family Caregiver: To minimize the burden to families, we have chosen a Treatment-as-Usual (TAU) comparison condition, where patients will receive their normal standard of care. Both study arms will receive palliative (specialized medical) care information at enrollment and complete questionnaires before and after the intervention or TAU period. Current practice for minors with life-limiting illnesses is to defer initial discussions of advanced care planning (pACP) until a medical crisis, so this is what the TAU control arm condition will consist of.
- FACE-Rare Intervention-Family Caregiver: FACE-Rare is a behavioral intervention that combines the CSNAT Pediatric Approach and the Respecting Choices® Next Steps ACP over 3 sessions.
  Sessions 1&2: CSNAT is an evidence-based process of family caregiver assessment and support in specialized medical (palliative) care. The CSNAT tool is structured around 16 categories of family caregiver support. With the goal to decrease caregiver burden, this process consists of 5 stages wherein a nurse or practitioner works with the caregiver to create a shared support plan for the child.
  Session 3: Respecting Choices® Next Steps- This advanced care planning (pACP) conversation engages families in a process for how to make future medical decisions
Arm/Group | FACE-Rare Intervention-Children | Treatment-as-Usual (TAU) Control- Children | FACE-Rare Intervention-Family Caregiver | TAU-control-Family Caregiver
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12 | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12 | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 0/9 | 0/12 | 0/9 | 0/12

LIMITATIONS AND CAVEATS:
Small sample size increased the risk of Type II error. We did not have enough power to detect differences in most of the outcome measures. Single site limits generalizability. Social desirability bias could have occurred with remote, but face-to-face, administration of study questionnaires.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT04855734/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT04855734/ICF_001.pdf